CLINICAL TRIAL: NCT01881100
Title: Randomized Clinical Trial on Resin Infiltration Versus Fluoride Varnish Treatment of Early Smooth-surface Caries Lesions in Deciduous Teeth
Brief Title: Randomized Trial on Resin Infiltration in Deciduous Teeth
Acronym: infiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Anna Turska Szybka, Phd,MD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No sponsor ID; WarsawMU (Other: WarsawMU)
Record Dates: First submitted 2013-06-16; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: White Spot Lesions; Caries
Keywords: resin infiltration; randomized clinical trial; fluoride varnish; caries lesion; deciduous teeth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- resin infiltration (Experimental): The test group (41 children) had caries lesions treated with the infiltration technique using Icon (DMG, Hamburg, Germany) and fluoride varnish (Duraphat, Colgate Palmolive, Hamburg, Germany)at baseline evaluation. Fluoride varnish was applied every control visit every three months during 1 year.
  Interventions: Other: resin infiltration; Other: fluoride varnish
- fluoride varnish (Active Comparator): The control group (40 children) had all tooth surfaces including WSL treated with fluoride varnish (Duraphat Colgate Palmolive, Hamburg, Germany)only at baseline evaluation and every control visit every three months during 1 year.
  Interventions: Other: fluoride varnish

INTERVENTIONS:
Other: resin infiltration — The test group (41 children) had caries lesions treated with the resin infiltration technique using Icon by the following procedure: rubber dam applying; etching with 15% hydrochloric acid for 120 s; surface rinsing and drying; dehydrating with ethanol for 30 s and air-drying; infiltrant resin infiltration with a syringe for 180 s; resin polymerization (polymerized by blue light - wavelength of 450 nm and intensity of 800mW/cm2; resin reapplication for 60 s and polymerization; rubber dam removal, and working on the infiltrated lesion with polishing rubbers. After the procedure fluoride varnish was applied.
  Other Names: Icon DMG Germany; Duraphat Colgate Palmolive Germany
  Arms: resin infiltration
Other: fluoride varnish — All tooth surfaces including WSL treated with fluoride varnish (2,26% F, Duraphat ® Colgate Palmolive, Hamburg, Germany).
  Other Names: Duraphat Colgate Palmolive, Hamburg, Germany

SUMMARY:
It was hypothesized that resin infiltration in conjunction with fluoride varnish treatment of smooth-surface caries lesions in deciduous teeth reduce considerably the progression of treated caries lesions, compared to fluoride varnish therapy only.

DETAILED DESCRIPTION:
* To determine the number of patients, sample size was based on data from studies assessing fluoride varnish efficacy in children with deciduous teeth (progression of caries reduction by 33 %)(95% CI, from 19 to 48%, P<0.0001); (α = 0.05; power = 80%; chi-square test2). The calculated sample size was 60 children and 120 white spot lesions. The initially planned number of participants was increased by expected 20% drop-out after 1 year, at least 72 children; the minimal number of treated active caries lesions amounted to 144.
* Participants were allocated to the "test" and to the "control" group, respectively, by computer-generated randomly permuted blocks using package blockrand in R statistical software, sealed in envelopes.
* The children were re-examined clinically by the same 2 examiners as at baseline evaluation.
* Statistical analyses were performed using statistical software STATISTICA 10 (StatSoft), the level of significance was set at 0.05. Intra-examiner reliability was assessed by kappa statistics.
* To compare average values between two independent groups U Mann-Whitney test was used (for e.g. to compare experimental group with the control one); Wilcoxon signed-rank test was used for paired samples (for e.g. to compare first measurement with final measurement for experimental group). Comparison of fractions was conducted using Pearson's chi-square test of independence and Z test. The 95% confidence intervals were calculated on the basis of normal approximation.

ELIGIBILITY:
Inclusion Criteria:

* at least two active smooth-surface caries lesions in deciduous teeth (ICDAS II code 2)
* a written consent of parents/ guardians for participation in the research study

Exclusion Criteria:

* age above 5.9 years
* systematic disease
* cavitated lesions
* enamel defects
* current participation in another study
* a planned change of residence within one year

Ages: 18 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Resin infiltration in conjunction with fluoride varnish treatment of smooth-surface caries lesions in deciduous teeth versus fluoride varnish therapy only. | one year
  The condition of treated white spot lesions (WSL) were scored using the Nyvad et al. system (17): I-WSL (Inactive WSL) - inactive spot lesion, when surface was becoming smooth, hard and glossy; S -WSL (Sound WSL) - invisible spot lesion taking the appearance of healthy enamel with proper translucency level and surface texture. Active enamel lesions and assessment scores 3-6 according to ICDAS II within a year were considered as decayed (D-Enamel/Dental cavity). Treatment was considered successful when lesions did not progress (I-WSL or S-WSL); unsuccessful when lesions remained active and enamel underwent erosion - i.e. caries occurred (D).

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Olczak-Kowalczyk, Ass. Prof., Study Director — Warsaw Medical University, 61 Żwirki i Wigury St.,02-091Warsaw; Dorota Olczak-Kowalczyk, Ass.Prof., Study Director — Warsaw Medical University, Poland
Locations (1):
- Dorota Olczak-Kowalczyk, Warsaw, Warsaw, 18 Miodowa Saint, Poland